CLINICAL TRIAL: NCT04766723
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial With an Open-label Period to Investigate the Efficacy and Safety of NT 201 in the Unilateral and Bilateral Treatment of Essential Tremor of the Upper Limb
Brief Title: A Study to Investigate the Efficacy and Safety of NT 201 (Botulinum Toxin) Compared With Placebo for the Treatment of Adult Participants With Essential Tremor in the Arm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011069; 2021-001988-24 (EudraCT Number)
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Essential Tremor of the Upper Limb
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT 201 (IncobotulinumtoxinA, Xeomin) (Experimental): Unilateral Treatment Period (1 treatment cycle): subjects to receive unilateral intramuscular injection of NT 201 (130-165 units) into muscles of the upper limb.
  Open Label Bilateral Treatment Period (1 treatment cycle): subjects to receive bilateral intramuscular injection of NT 201 (130-165 units) into muscles of the upper limbs.
  Interventions: Drug: NT 201
- Placebo (Placebo Comparator): Unilateral Treatment Period (1 treatment cycle): subjects to receive unilateral intramuscular placebo injection into muscles of the upper limb.
  Open Label Bilateral Treatment Period (1 treatment cycle): subjects to receive bilateral intramuscular injection of NT 201 (130-165 units per arm) into muscles of the upper limbs.
  Interventions: Drug: NT 201; Drug: Placebo

INTERVENTIONS:
Drug: NT 201 — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: Incobotulinumtoxin A; IncobotulinumtoxinA; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a single treatment with administration of NT 201 (botulinum toxin) is superior to placebo (no medicine) for one-sided treatment of essential tremor in the arm (Unilateral Period). Participants will be assigned to the treatment groups by chance and neither the participants nor the research staff who interact with them will know the allocation.

The following treatment cycle will investigate the safety and tolerability of two-sided treatment with NT 201 (botulinum toxin) (Open Label Bliaterial Period). All participants will receive NT 201 treatment.

ELIGIBILITY:
Inclusion Criteria:

- Score of ≥ 2 (at least 1 cm tremor amplitude) in at least two out of three maneuvers of test item 4 (upper limb tremor) confirmed by an independent TETRAS expert by means of video assessment.

Exclusion Criteria:

* History or presence of day-to-day fluctuations in ET which would jeopardize meaningful tremor assessment over time, e.g. severe tremor on one day and minimal or no tremor on another day.
* Other neurological signs, such as dystonia, ataxia, or parkinsonism, which in the judgment of the investigator could interfere with the ET diagnosis and/or assessment of ET in ULs.
* Tremor types other than ET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Change from study baseline to Week 6 in maximum tremor amplitude measurement at wrist level during the unilateral treatment period | From baseline to week 6

SECONDARY OUTCOMES:
Change from study baseline to Week 6 in the Essential Tremor Rating Assessment Scale [TETRAS] Performance dominant upper limb [UL] score | From baseline to week 6
Change from study baseline to Week 6 in TETRAS Activities of Daily Living [ADL] UL score | From baseline to week 6
Change from study baseline to Week 6 in TETRAS ADL Functional Impact score | From baseline to week 6
Subject´s Global Impression of Change Scale [GICS] score of motor dominant UL at Week 6 | Week 6
Investigator´s Global Impression of Change Scale [GICS] score of motor dominant UL at Week 6 | Week 6
Change from Cycle 2 baseline to Week 6 in TETRAS Performance dominant UL score | Week 24 to week 36
Change from Cycle 2 baseline to Week 6 in TETRAS Performance subscale score | Week 24 to week 36
Change from Cycle 2 baseline to Week 6 in TETRAS ADL UL score | Week 24 to week 36
Change from Cycle 2 baseline to Week 6 in TETRAS ADL Functional Impact score | Week 24 to week 36
Incidence of treatment-emergent AEs [TEAEs] related to treatment | From baseline to week 36

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (14):
- United States (9):
  - USF, Department of Neurology, Merz Investigational Site #0010020, Tampa, Florida
  - University of Nebraska Medical Center, Merz Investigational Site #0010269, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Merz Investigational Site #0010457, Las Vegas, Nevada
  - Mount Sinai Medical Center, Merz Investigational Site #0010191, New York, New York
  - Vanderbilt University Medical Center, Neuroscience Institute, Merz Investigational Site #0010206, Nashville, Tennessee
  - Houston Methodist Neurological Institute, Merz Investigational Site #0010226, Houston, Texas
  - Medstar Georgetown Neurology, Merz Investigational Site #0010231, McLean, Virginia
  - UW Medical Center - Montlake, Merz Investigational Site #0010450, Seattle, Washington
  - Selkirk Neurology, Merz Investigational Site #0010456, Spokane, Washington
- London Health Sciences Centre, Merz Investigational Site #0010087, London, Ontario, Canada
- Poland (4):
  - Specjalistyczne Gabinety, Merz Investigational Site #0480059, Krakow
  - NeuroKlinika Gabinet Lekarski, Merz Investigational Site #0480101, Lodz
  - Instytut Zdrowia Dr. Boczarska-Jedynak, Oświęcim
  - Mazowiecki Szpital Bródnowski, Merz Investigational Site #0480064, Warsaw

IPD SHARING:
Plan to Share IPD: No